CLINICAL TRIAL: NCT04205773
Title: Confirmation of Epidural Catheter Location by Epidural Pressure Waveform Recordings by the CompuFlo Epidural Instrument
Brief Title: Epidural Catheter Location by Epidural Pressure Waveform
Status: Completed | Type: Observational
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Other Study IDs: EESOA3
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CompuFlo — After priming with 5 mL saline, the catheter was connected to CompuFlo to record the occurrence of pulsatile waveforms and/or their disappearance during its removal

SUMMARY:
The aim of this preliminary study was to evaluate the new CompuFlo instrument which allows pulsatile waveform recordings.

DETAILED DESCRIPTION:
30 epidural catheters previously successfully used for obstetric anesthesia or analgesia and about to be removed were tested. All patients were given 5 mL 2% lidocaine to test the catheter before its removal. After priming with 5 mL saline, the catheter was connected to CompuFlo to record the occurrence of pulsatile waveforms and/or their disappearance during its removal. The epidural catheter was marked at the skin level to record the distance between the skin at the time of measurements. The power analysis required a sample of 30 observations to set 80% test power and 95% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients
* Must have an epidural catheter

Exclusion criteria

• Non-obstetric patients

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant patients
Study Population: Obstetric patients who received an epidural block and have an epidural catheter
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
pulsatile waveforms observation (presence or absence) | 30 minutes
  The epidural catheter was considered to be in the epidural space if the appearance of pulsatile waveforms were observed, and confirmed by the occurrence of L2-3 sensory block after the test dose. The disappearance of the pulsatile waveforms when the catheter was extracted from the epidural space was also noted.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (2):
- Italy (2):
  - EESOA Maternal Neonatal Simulation Centre, Roma
  - Città di Roma Hospital, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Capogna G, Coccoluto A, Capogna E, Del Vecchio A. Objective Evaluation of a New Epidural Simulator by the CompuFlo(R) Epidural Instrument. Anesthesiol Res Pract. 2018 Jun 26;2018:4710263. doi: 10.1155/2018/4710263. eCollection 2018. PMID 30046305